CLINICAL TRIAL: NCT01884610
Title: Multi Centre Controlled Study on the Impact of Stem Cell Donation Either After Mobilisation With Granulocyte Colony Stimulating Factor or Bone Marrow Harvest on Unrelated Bone Marrow Donors.
Brief Title: Study on the Impact of Stem Cell Donation and Bone Marrow Harvesting on Unrelated Donors
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: British Bone Marrow Registry (Unknown); Anthony Nolan Research Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: BRD/06/143
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Chromosome Aberrations
MeSH Terms: conditions — Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fixed ( methanol/acetic acid ) chromosome preparations solution and genomic DNA.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Granulocyte Colony Stimulating Factor (GCSF) is used extensively as a means of mobilising donor peripheral blood stem cells as an alternative to bone marrow harvesting for the purpose of recipient stem cell transplantation. The principal objective of the research is to study any longterm genetic effects of GCSF in the peripheral blood white cells of unrelated blood stem cell donors.

The study subjects will be Retrospective and Prospective voluntary unrelated donors on the Anthony Nolan Bone Marrow Registry being harvested at the Royal Free Hospital and University College Hospital, London and British Bone Marrow Registry donors harvested at the Royal Free Hospital and BUPA Glen Vale in Bristol.

All participants in the Prospective Arm will be asked to donate one 5-10ml sample of blood at study entry prior to stem cell donation and further samples at 120 and 360 days post donation. Those found to carry aneuploid cell clones at these time points will be asked for a further 5-10ml blood sample at least twice - at the end of 24 months and 36 months respectively. The Retrospective and Positive Control group will be asked to supply one 5-10ml sample of blood.

DETAILED DESCRIPTION:
The aim of this study is to detect any genetic differences between bone marrow and PBSC unrelated donors, post donation and confirm or refute the observations of "long-term genetic or epigenetic effects" published by Nagler et al[Nagler,A. et al. Exp.Haem (2004) 32;122-30]. The employment of more sensitive methods such as iFISH and gene array analysis to assess any permanent genetic changes, our primary objective, will make our study more robust.

There will be two arms:

i) Retrospective arm - the peripheral blood of unrelated donors who donated 3 to 5 years previously will be screened.

ii) Prospective arm - peripheral blood of unrelated donors will be examined prior to donation and at 120 and 360 day's post-donation. In those found to have aneuploid changes at these time points, there will be additional sampling at 24 and 36 months and if necessary these donors will be followed up.

Each arm of the study will include 50 BM unrelated donors and 50 PBSC unrelated donors giving a total sample population of around 200 unrelated donors. There will be one positive control group of 50 patients with a range of haematological malignancies. The blood samples taken from both BM and PBSC donors prior to donation will act as internal negative controls.

ELIGIBILITY:
Inclusion Criteria:

Donors of peripheral blood stem cells

Exclusion Criteria:

Relatives suffering from blood cancer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Donors of peripheral blood stem cells, who have agreed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Chromosome aberration in peripheral blood lymphocytes | 180 days
  Peripheral blood stem cells donors who have been administered GCSF are monitored for genetic damage. This is performed by screening samples of peripheral blood lymphocytes taken before and after GCSF administration (at day 0, day 90 and day 180) for chromosome aberrations using FISH (fluorescence in situ hybridisation) methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth P Nacheva, MD PhD FRCPath, Principal Investigator — University College London (UCL) Cancer Institute